CLINICAL TRIAL: NCT01832363
Title: Single-Session Bronchial Thermoplasty for Severe Asthmatics Guided by HXe MRI
Brief Title: Bronchial Thermoplasty for Severe Asthmatics Guided by HXe MRI
Acronym: HXe-BT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xemed LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Washington University School of Medicine (Other); University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MagniXene-112397; R44HL112397 (NIH)
Record Dates: First submitted 2013-03-28; First posted 2013-04-16 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-01

CONDITIONS: Asthma
Keywords: Severe asthma; Bronchial thermoplasty; MagniXene; Hyperpolarized Xenon; HXe; HyXe
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HXe MRI guided treatment sequence for BT (Experimental): Patients in this arm will undergo bronchial thermoplasty treatment where the first session of the procedure will target the six most problematic airways as determined with HXe imaging. Patients will have the remaining of the airways treated in the two subsequent sessions.
  Interventions: Drug: HXe MRI guided treatment sequence for BT
- Standard treatment sequence for BT (control) (Active Comparator): Patients in this arm will undergo standard treatment sequence of bronchial thermoplasty. To preserve the blind of the procedure to the subjects, the same timeline and clinical measures will be followed as for HXe guided patients.
  Interventions: Other: Standard treatment sequence for BT (control)

INTERVENTIONS:
Drug: HXe MRI guided treatment sequence for BT — HXe MRI consists in imaging the inhaled xenon gas inside the human lungs during a short breath-hold. High resolution 3D maps of the HXe distribution inside the lungs provide information regarding ventilation of the lungs, as the signal is proportional to the local concentration of HXe. A high MRI signal translates in unobstructed ventilation, while ventilation defects appear as dark regions on the map. HXe MRI will be performed pre and post bronchodilator in order to determine the airways which potentially are the most responsive to BT treatment. All HXe MRI images will be repeated within the same day for consistency check and after three weeks to study temporal variability. The reactivity of the airways will establish the treatment order, with the most problematic airways to be treated in the first BT session (not to exceed six).
  Other Names: MagniXene; Hyperpolarized Xenon; HXe
  Arms: HXe MRI guided treatment sequence for BT
Other: Standard treatment sequence for BT (control) — Patients undergoing standard BT procedure will have HXe MRI performed at time intervals similar to HXe MRI guided BT patients. While HXe images will not be used for guiding the sequence for airways to receive the BT treatment, metrics extracted from HXe images will be compared with clinically accepted asthma severity metrics (spirometry and asthma questionnaires) to assess HXe MRI as a biomarker for asthma severity.
  Other Names: MagniXene; Hyperpolarized Xenon; HXe
  Arms: Standard treatment sequence for BT (control)

SUMMARY:
The purpose of this study is to determine if the bronchial thermoplasty treatment can be guided through hyperpolarized xenon lung MRI.

DETAILED DESCRIPTION:
This study explores the feasibility of using hyperpolarized xenon (HXe) Magnetic Resonance Imaging (MRI) as a diagnostic imaging agent to prioritize the order of airway treatment by bronchial thermoplasty, rather than the FDA approved pre-established treatment sequence that is performed today.

The Alair® Bronchial Thermoplasty System is an FDA approved device clinically proven to be effective in treating severe asthma patients who are not well controlled with inhaled corticosteroids and long acting beta agonists. Bronchial thermoplasty (BT) is a procedure that reduces excessive airway smooth muscle by radio wave ablation, thus decreasing the ability of the airways to constrict during an asthma attack. The BT procedure is performed in three separate outpatient treatment sessions, each treating pre-established regions of the lungs. The sessions are separated by at least three weeks healing time.

MagniXene® is pure xenon gas which is magnetically altered to become a contrast agent for magnetic resonance imaging of the lungs. The subject inhales the hyperpolarized xenon while inside the MRI scanner and a highly detailed ventilation map of the lung spaces is acquired during a short breath-hold. By detecting unventilated regions and airway reactivity using HXe images, a prioritized scheme for performing bronchial thermoplasty can be elaborated to treat the most problematic airways within the first BT session. In this study the rest of the airway will be treated in the following two sessions, such that all the airways are treated in the end as in the standard procedure.

This study will include approximately 30 patients clinically indicated to undergo bronchial thermoplasty. Half of the patients will be randomly assigned to receive HXe guided BT, while the other half will receive standard BT procedure. HXe images and clinical measures of asthma disease severity, such as Asthma Quality of Life Questionnaire (AQLQ), Asthma Control Test (ACT), morning expiratory peak flow (AM-PEF), pulmonary function tests (PFT), will be acquired at three time points interleaved with the BT sessions: before BT, 12 weeks after first session of BT, and 12 weeks after the third session of BT (approximately 36 weeks from baseline). HXe MRI will be repeated within the same day after bronchodilator treatment of the patient to establish airways reactivity. Additionally, a three-week follow up for HXe MRI will allow us to study temporal variability of HXe metrics. A total of six HXe imaging sessions (distinctive days), each including at least four HXe images will be dedicated to each patient.

The primary outcome of this study will be to determine whether the standard full BT treatment is superior to a single session guided treatment. The statistical metric will be the incremental change in the AQLQ score.

ELIGIBILITY:
Inclusion Criteria (bronchial thermoplasty):

* Males or females age 18 or greater and less than 65.
* Subject has asthma and is taking regular maintenance medication for past 12 months that includes:

  * Inhaled corticosteroid (ICS) at a dosage greater than 1000μg beclomethasone per day or equivalent, AND long acting ß2-agonist (LABA) at a dosage of ≥100μg per day Salmeterol or equivalent.
  * Other asthma medications such as leukotriene modifiers, or anti-immunoglobulin E (IgE), are acceptable (Subjects on Xolair® must have been on Xolair for greater than 1 year).
* Asthma confirmed by: (a) b-agonist reversibility of FEV1 ≥ 12 % following 360mcg albuterol OR (b) 20% fall in forced expiratory volume in 1 second (PC20-FEV1) after a challenge with methacholine ≤ 8 mg/ml if not receiving an inhaled corticosteroid (ICS) or ≤ 16 mg/ml if receiving an ICS.
* FEV1 ≥ 50% predicted pre-bronchodilator.
* Asthma symptoms on at least two days or one night per week over the last 2 weeks.
* Subject is a non-smoker for 1 year or greater (if former smoker, less than 10 pack-years total smoking history).
* Patient has a clinical indication for bronchial thermoplasty as decided by their treating physician.
* Ability to undergo bronchoscopy in the opinion of the investigator.

Exclusion Criteria (bronchial thermoplasty):

* Asthma exacerbation (ED visit, hospitalization, course of increased systemic steroids, or urgent health care visit for asthma) during the prior four weeks.
* Asthma exacerbation requiring hospitalization during the prior six weeks.
* Chronic oral steroid therapy greater than 30 mg per day.
* Respiratory tract infection within past 4 weeks
* Subject has a known sensitivity to medications required to perform bronchoscopy (such as lidocaine, atropine and benzodiazepines).
* Subject is undergoing immunosuppressant therapy (e.g., methotrexate).
* Subject is on anticoagulant medication.
* Subject has bleeding diathesis, platelet dysfunction, and thrombocytopenia with platelet count less than 125,000/mm2 or known coagulopathy (INR > 1.5).
* Subject has other respiratory diseases including interstitial lung disease, emphysema, cystic fibrosis, vocal cord dysfunction, mechanical upper airway obstruction, untreated obstructive sleep apnea, Churg-Strauss syndrome, cardiac dysfunction, and allergic bronchopulmonary aspergillosis (total IgE of >1000 Units/mL with positive specific IgE to aspergillus and evidence of central bronchiectasis).
* Subject has segmental atelectasis, lobar consolidation, significant or unstable pulmonary infiltrate, or pneumothorax, confirmed on x-ray.
* Subject has clinically significant cardiovascular disease, including myocardial infarction, angina, cardiac dysrhythmia, conduction defect, cardiomyopathy, aortic aneurysm, or stroke.
* Subject has uncontrolled hypertension (>200mm Hg systolic or >100mm Hg diastolic pressure).
* Subject uses an internal or external pacemaker or cardiac defibrillator.
* Chronic diseases (other than asthma) that in the opinion of the investigator would prevent participation in the trial or put the participant at risk by participation, e.g. chronic diseases of the lung (other than asthma), heart, liver, kidney, or nervous system, or immunodeficiency
* History of cigarette smoking with > 10 pack years total
* Use of investigative drugs or intervention trials in the 30 days prior to enrollment or during the duration of the study
* Any condition or compliance issue which in the opinion of the investigator might interfere with participation in the study

Exclusion Criteria (Magnetic Resonance Imaging):

* Obesity exceeding the scanner capability
* Metal implants or non-removable metal piercings
* Inability to tolerate MRI scanning due to claustrophobia

Exclusion Criteria (HXe inhalation):

* Pregnancy or intention to become pregnant
* Neurological or cardiac comorbidities
* Hemoglobin level below 10 g/dl as determined in a recent (within 12 months) measurement

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Change in Asthma Quality of Life Questionnaire (AQLQ) from baseline | 2.5 years
  Asthma Quality of Life Questionnaire (AQLQ) is the primary outcome of this study. We will test whether the standard (unguided) three session BT treatment is superior to the a HXe MRI guided, single session BT treatment. There will be three time points of measure of the AQLQ score: before the BT session (baseline), 12 weeks after the first BT session, and 12 weeks after the third (last) BT session (approximately 36 weeks from baseline).

SECONDARY OUTCOMES:
Assessment of HXe MRI as an imaging biomarker for asthma disease severity | 2.5 years
  HXe MRI data analysis can quantify measures of lung functionality such as fractional ventilation (V) and bronchodilator response (BD), as well as temporal variability of these metrics (dV and dBD). These measures will be compared against existing clinical parameters defining asthma disease severity, such as questionnaire scores: AQLQ and Asthma Control Test; as well as spirometry measures: Forced Expiratory Volume in one second (FEV1), and morning Peak Expiratory Flow (AM-PEF), in search for correlations and to demonstrate that HXe can be considered a clinical measure for asthma disease severity.

CONTACTS AND LOCATIONS:
Overall Officials: Iulian C Ruset, PhD, Principal Investigator — Xemed LLC; James Quirk, PhD, Principal Investigator — Washington University School of Medicine; Nicholas Tustison, PhD, Principal Investigator — University of Virginia
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States